CLINICAL TRIAL: NCT06166056
Title: A Randomised, Double-blind, Placebo-controlled Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Inhaled CHF6333 After Single Ascending Doses in Healthy Volunteers and One Single Dose in Adult Subjects With Bronchiectasis, Followed by a Placebo-controlled, Repeated Dose, 3-way Cross-over in Adult Subjects With Bronchiectasis
Brief Title: A Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Inhaled CHF6333 After Single Doses in Healthy Volunteers and After Single and Repeated Doses in Subjects With Bronchiectasis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLI-06333CA1-01
Record Dates: First submitted 2023-11-22; First posted 2023-12-12 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Intervention Model Description: Part I: randomised, double-blind, placebo-controlled, single ascending dose, alternating cross-over design in HV and single dose in subjects with BE. Part II: randomised, double-blind, placebo-controlled, repeated-dose, 3-way cross-over design in subjects with BE.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: CHF6333 (Experimental): CHF6333 active (Part I - SAD): once daily inhaled single dose of CHF6333 at each period (three dose levels for HVs and one dose level for BE subjects).
  CHF6333 active (Part II - MD): once daily inhaled multiple dose of CHF6333 for 28 days consecutive days (two dose levels for BE subjects).
  Interventions: Drug: CHF6333
- Placebo comparator: CHF6333 Placebo (Placebo Comparator): CHF6333 placebo (Part I - SAD): once daily inhaled single dose of placebo matching CHF6333 at each period.
  CHF6333 placebo (Part II - MD): once daily inhaled multiple dose of placebo matching CHF6333 for 28 days consecutive days.
  Interventions: Drug: CHF6333 Placebo

INTERVENTIONS:
Drug: CHF6333 — CHF6333 Part I SAD; CHF6333 Part II MD.
  Arms: Experimental: CHF6333
Drug: CHF6333 Placebo — Placebo Part I SAD; Placebo Part II MD.
  Arms: Placebo comparator: CHF6333 Placebo

SUMMARY:
The aim of this clinical trial is to assess the safety of:

* single doses of the study drug CHF6333 in Healthy Volunteers (HVs) and in subjects with Bronchiectasis (BE) - Part I
* repeated doses of the study drug CHF6333 in subjects with BE - Part II

ELIGIBILITY:
HV Inclusion Criteria:

1. Signed and dated informed consent obtained prior to any study-related procedure;
2. Healthy male or female subject ≥18 and ≤60 years of age at screening;
3. Ability to understand the study procedures and the risks involved, and to be trained to use inhalers correctly and to generate sufficient peak inspiratory flow (PIF) (at least 40 L/min) using the In-Check Dial set as per "GenuAir" inhaler resistance, at screening;
4. Body mass index (BMI) ≥18 and ≤35 kg/m2 at screening;
5. Non-smokers or ex-smokers who smoked <5 pack-years and stopped smoking >1 year prior to screening;
6. Good physical and mental status, determined via assessment of medical history and clinical examination, at screening and prior to randomisation;
7. Vital signs within normal limits at screening and prior to randomisation: diastolic blood pressure (DBP) ≥40 and ≤89 mmHg, and systolic blood pressure (SBP) ≥90 and ≤139 mmHg; body temperature <37.5°C;
8. Triplicate 12-lead electrocardiogram (ECG) considered as normal (40 ≤ heart rate ≤110 bpm, 120 ms ≤ PR ≤210 ms, QRS ≤120 ms, Fridericia corrected QT interval [QTcF] ≤450 ms for males and QTcF ≤470 ms for females) at screening and prior to randomisation;
9. Lung function measurements within limits at screening and prior to randomisation: forced expiratory volume in 1 second (FEV1) >80% predicted and FEV1/forced vital capacity (FVC) ratio >0.70;
10. Male subjects willing to use a male condom throughout the study if they have women of childbearing potential (WOCBP) partners; male subjects with non-WOCBP partners or who are sterile do not have contraception requirements;
11. Female subjects (if WOCBP) and/or their partners (if fertile) must be willing to use a highly effective birth control method, preferably with low user dependency, throughout the study; female subjects who are non-WOCBP or who have non-fertile partners do not have contraception requirements.

HV Exclusion Criteria:

1. Participation in another clinical study where investigational drug was received and the last investigations were performed less than 3 months prior to randomisation;
2. Clinically relevant and uncontrolled respiratory, cardiac, hepatic, gastrointestinal, renal, endocrine, hematologic, metabolic, neurological, or psychiatric disorders that may interfere with successful completion of this protocol, according to the investigator's judgment;
3. Clinically relevant abnormal laboratory values at screening suggesting an unknown disease and requiring further clinical investigation or which may impact the safety of the subject or the evaluation of the results of the study, according to the investigator's judgment;
4. History of respiratory diseases;
5. Positive human immunodeficiency virus (HIV) 1 or HIV2 serology results at screening;
6. Hepatitis serology results which indicate acute or chronic hepatitis B (HB) or hepatitis C virus (HCV) at screening;
7. Documented coronavirus disease 2019 (COVID-19) diagnosis within 2 weeks prior to screening or prior to randomisation, or associated complications/symptoms, which have not resolved within 2 weeks prior to screening;
8. Blood donation or blood loss (equal or more than 450 mL) less than 2 months prior to screening or prior to randomisation;
9. Abnormal liver enzymes at screening or prior to randomisation (alanine aminotransferase [ALT] or aspartate aminotransferase [AST] or bilirubin: >1.5× upper limit of normal [ULN]);
10. Positive urine test for cotinine at screening or prior to randomisation;
11. Documented history of alcohol abuse within 12 months prior to screening or a positive alcohol breath test at screening or prior to randomisation;
12. Documented history of drug abuse within 12 months prior to screening or a positive urine drug screen at screening or prior to randomisation;
13. Treatment with prohibited concomitant medications or if the subject is expected to take prohibited concomitant medications during the study;
14. Presence of any current infection, or previous infection that resolved less than 7 days prior to screening or prior to randomisation;
15. Known intolerance and/or hypersensitivity to any of the excipients contained in the formulation used in the study;
16. Unsuitable veins for repeated venepuncture;
17. Heavy caffeine drinker;
18. For females only: pregnant or lactating women, where pregnancy is defined as the state of a female after conception and until termination of the gestation, confirmed by a positive serum human chorionic gonadotropin laboratory test. A serum pregnancy test is to be performed at screening and a urine pregnancy test is to be performed prior to randomisation;
19. Use of any kind of electronic smoking devices within 6 months prior to screening.

Part I BE subjects Inclusion Criteria:

1. Signed and dated informed consent obtained prior to any study-related procedure;
2. Male or female subject ≥18 and ≤80 years of age at screening;
3. Clinical history consistent with BE (cough, chronic sputum production, and/or recurrent respiratory infections) that is confirmed by chest computed tomography (CT) demonstrating BE affecting 1 or more lobes (confirmation may be based on prior chest CT); subjects whose past chest radiographic image records or report are not available will undergo chest CT scan during screening;
4. Post-bronchodilator FEV1 ≥50% of the predicted value at screening;
5. If currently receiving treatment for BE, this treatment should be administered at a stable dose;
6. Subjects in a stable clinical condition with no exacerbation of BE for at least 4 weeks prior to randomisation. A pulmonary exacerbation is defined as a deterioration in three or more of the key symptoms for at least 48 hours (cough, sputum volume and/or consistency, sputum purulence, breathlessness and/or exercise tolerance, fatigue and/or malaise, haemoptysis) AND a clinician-prescribed course of antibiotics;
7. Vital signs within normal limits at screening and prior to randomisation: DBP ≥40 and ≤89 mmHg, and SBP ≥90 and ≤150 mmHg; body temperature <37.5°C;
8. Ability to understand the study procedures and the risks involved, and the ability to be trained to use the inhalers correctly and to generate sufficient PIF (at least 40 L/min) using the In-Check Dial set as per "GenuAir" inhaler resistance, at screening;
9. Male subjects willing to use a male condom throughout the study if they have WOCBP partners; male subjects with non-WOCBP partners or who are sterile do not have contraception requirements;
10. Female subjects (if WOCBP) and/or their partners (if fertile) must be willing to use a highly effective birth control method, preferably with low user dependency, throughout the study; female subjects who are non-WOCBP or who have non-fertile partners do not have contraception requirements.

Part I BE subjects Exclusion Criteria:

1. History of a clinically meaningful unstable or uncontrolled chronic comorbidity that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering the study drug to the subject;
2. Acute symptomatic respiratory tract infection which constitutes an increase from the subject's baseline, per the investigator's judgment, within 4 weeks prior to randomisation;
3. Abnormal and clinically significant 12-lead ECG at screening or prior to randomisation that results in an active medical problem, which may impact the safety of the subject, per the investigator's judgment. Male subjects with QTcF >450 ms and female subjects with QTcF >470 ms cannot be enrolled;
4. Clinically significant abnormal laboratory values at screening that, in the opinion of the investigator, may put the subject at risk by participating in the study, or interfere with the subject's treatment or assessment, or influence the results of the study;
5. Participation in another clinical study, where investigational drug was received less than 30 days or less than 5 half-lives of the previous administered product (whichever is longer) prior to screening; participation in another clinical study is also not allowed between screening and randomisation;
6. Primary diagnosis of asthma, as determined by the investigator;
7. Concomitant diagnosis of cystic fibrosis;
8. Diagnosis of chronic obstructive pulmonary disease (COPD) made by a clinician, with airflow obstruction (post-bronchodilator FEV1/FVC ratio <0.7) and at least a 10 pack-year smoking history; subjects with documented COPD but without airflow obstruction or smoking history will be permitted;
9. Current smokers; ex-smokers must have stopped for at least 1 year prior to screening (≥6 months for electronic smoking devices);
10. Subjects with an active tuberculous mycobacteria (TM) or non-tuberculous mycobacteria (NTM) infection requiring or receiving antibiotic treatment, an active allergic bronchopulmonary aspergillosis requiring treatment with corticosteroids or anti-fungal therapy, and/or a connective tissue disease (CTD) receiving an immunosuppressive treatment equivalent to >10 mg prednisolone daily or systemic immunosuppression;
11. Diagnosis of common variable immunodeficiency (CVID) or other immunodeficiencies requiring immunoglobulin treatment, based on subject history;
12. Diagnosis of rheumatoid arthritis;
13. Malignancy that has not been in complete remission for at least 1 year or any untreated localised carcinomas;
14. History of solid organ/haematological transplantation and receiving immunosuppressive therapy;
15. Use of any antimicrobials (oral, inhaled, or intravenous) within 4 weeks prior to randomisation, except for subjects who are on stable treatment with macrolide antibiotics (for at least 3 months);
16. Medical history of discontinuation of previous inhaled therapy due to bronchospasm or intolerance;
17. Documented COVID-19 diagnosis within 4 weeks prior to randomisation, or associated complications/symptoms;
18. Diagnosis of alpha-1-antitrypsin (AAT) deficiency defined as an AAT serum level <110 mg/dL; a prior test result of AAT serum level to confirm the diagnosis will be acceptable. In the event that a prior result is not available, a new test will be performed during the screening period and the result considered for the eligibility at randomisation.
19. Treatment with prohibited concomitant medications or if the subject is expected to take prohibited concomitant medications during the study;
20. Subjects treated with monoclonal antibodies (mAbs) for any respiratory conditions;
21. Subjects with traction BE;
22. For females only: pregnant or lactating women, where pregnancy is defined as the state of a female after conception and until termination of the gestation, confirmed by a positive serum human chorionic gonadotropin laboratory test. A serum pregnancy test is to be performed at screening, and a urine pregnancy test is to be performed prior to randomisation;
23. Positive HIV1 or HIV2 serology results at screening;
24. Hepatitis serology results which indicate acute or chronic HB or HCV at screening;
25. BMI ≤17 kg/m2 at screening.

Part II BE subjects Inclusion Criteria: the subjects must meet all the inclusion criteria listed in Part I for subjects with BE (Cohort B), except the inclusion criterion below:

4. Post-bronchodilator FEV1 ≥30% of the predicted value at screening.

The subjects must also meet the additional inclusion criteria listed below:

11. Subjects who are regular daily sputum producers and who are able to provide at least one sputum sample at screening and two sputum samples prior to randomisation; 12. Subjects with active NE level in sputum sample at screening, defined by either a positive bacterial culture in a local laboratory (a positive result for any pathogen will be accepted for eligibility) or by a positive reading of the NEATstik® in vitro diagnostic test.

Part II BE subjects Exclusion Criteria:

See the list of criteria in Part I for subjects with BE (Cohort B), except the exclusion criterion below:

15. Use of oral or inhaled antibiotics < 3 months prior to randomization as chronic treatment for BE. Patients on antibiotics as chronic treatment should have been on such treatment for ≥ 3 months prior to randomization while meeting all other inclusion and exclusion criteria.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of single ascending doses of CHF6333 in HVs and a single dose in subjects with BE (Part I), and repeated doses in subjects with BE (Part II), in terms of AEs | Through study completion. Part I: an average of 12 weeks and 8 weeks respectively for HVs and BE subjects. Part II: an avarage of 26 weeks
Safety and tolerability of single ascending doses of CHF6333 in HVs and a single dose in subjects with BE (Part I), and repeated doses in subjects with BE (Part II), in terms of vital signs | Part I:screening, day(D)-1, D1(from pre-dose until 96hrs post-dose HV, 6hrs post-dose BE), 14 to 21D post-dose.Part II:screening, D-1, D1 and 27(from pre-dose until 6hrs post-dose), D28(from pre-dose until 2hrs post-dose), 14 to 21D after last dose
  Arterial blood pressure (SBP and DBP)
heart rate (HR) | Part I: at day1 from pre-dose until 24hrs post-dose. Part II: at day1 and 27 from pre-dose until 8hrs post-dose
  Safety and tolerability of single ascending doses of CHF6333 in HVs and a single dose in subjects with BE (Part I), and repeated doses in subjects with BE (Part II).
Safety and tolerability of single ascending doses of CHF6333 in HVs and a single dose in subjects with BE (Part I), and repeated doses in subjects with BE (Part II), in terms of 12-Lead ECG parameters from Holter: PR interval | Part I: at day1 from pre-dose until 24hrs post-dose. Part II: at day1 and 27 from pre-dose until 8hrs post-dose
  Part I HVs only and Part II
Safety and tolerability of single ascending doses of CHF6333 in HVs and a single dose in subjects with BE (Part I), and repeated doses in subjects with BE (Part II), in terms of 12-Lead ECG parameters from Holter: QRS interval | Part I: at day1 from pre-dose until 24hrs post-dose. Part II: at day1 and 27 from pre-dose until 8hrs post-dose
  Part I HVs only and Part II
Safety and tolerability of single ascending doses of CHF6333 in HVs and a single dose in subjects with BE (Part I), and repeated doses in subjects with BE (Part II), in terms of 12-Lead ECG parameters from Holter: Fridericia-corrected QT interval (QTcF) | Part I: at day1 from pre-dose until 24hrs post-dose. Part II: at day1 and 27 from pre-dose until 8hrs post-dose
  Part I HVs only and Part II
Safety and tolerability of single ascending doses of CHF6333 in HVs and a single dose in subjects with BE (Part I), and repeated doses in subjects with BE (Part II), in terms of lung function parameters: FEV1 | Part I: screening, day-1, day1 (from pre-dose until 24hrs post-dose for HVs and 6hrs post-dose for BE. Part II: screening, day-1, day1 and 27 (from pre-dose until 6hrs post-dose), day 28 (from pre-dose until 2hrs post-dose
Safety and tolerability of single ascending doses of CHF6333 in HVs and a single dose in subjects with BE (Part I), and repeated doses in subjects with BE (Part II), in terms of lung function parameters: FVC | Part I: screening, day-1, day1 (from pre-dose until 24hrs post-dose for HVs and 6hrs post-dose for BE. Part II: screening, day-1, day1 and 27 (from pre-dose until 6hrs post-dose), day 28 (from pre-dose until 2hrs post-dose
Safety and tolerability of single ascending doses of CHF6333 in HVs and a single dose in subjects with BE (Part I), and repeated doses in subjects with BE (Part II), in terms of lung function parameters: FEV1/FVC ratio | Part I: screening, day-1, day1 (from pre-dose until 24hrs post-dose for HVs and 6hrs post-dose for BE. Part II: screening, day-1, day1 and 27 (from pre-dose until 6hrs post-dose), day 28 (from pre-dose until 2hrs post-dose
Safety and tolerability of single ascending doses of CHF6333 in HVs and a single dose in subjects with BE (Part I), and repeated doses in subjects with BE (Part II), in terms of lung function parameters: FEV1 percentage of predicted | Part I: screening, day-1, day1 (from pre-dose until 24hrs post-dose for HVs and 6hrs post-dose for BE. Part II: screening, day-1, day1 and 27 (from pre-dose until 6hrs post-dose), day 28 (from pre-dose until 2hrs post-dose
Number of participants with clinical laboratory tests: Haematology | Part I: screening, day-1 and day5 (pre-dose) for HVs/FU for BE. Part II: screening, day-1 and 27 (pre-dose)
  Safety and tolerability of single ascending doses of CHF6333 in HVs and a single dose in subjects with BE (Part I), and repeated doses in subjects with BE (Part II), in terms of clinical laboratory tests: Haematology
Number of participants with clinical laboratory tests: Biochemistry | Part I: screening, day-1 and day5 (pre-dose) for HVs/FU for BE. Part II: screening, day-1 and 27 (pre-dose)
  Safety and tolerability of single ascending doses of CHF6333 in HVs and a single dose in subjects with BE (Part I), and repeated doses in subjects with BE (Part II), in terms of clinical laboratory tests: Biochemistry
Number of participants with clinical laboratory tests: Urinalysis | Part I: screening, day-1 and day 5 (pre-dose) for HVs/FU for BE. Part II: screening, day-1 and 27 (pre-dose)
  Safety and tolerability of single ascending doses of CHF6333 in HVs and a single dose in subjects with BE (Part I), and repeated doses in subjects with BE (Part II), in terms of clinical laboratory tests: Urinalysis

SECONDARY OUTCOMES:
Pharmacokinetic variables in plasma in HVs only (Part I), in terms of Area Under the Curve | Day 1: from pre-dose until 96 hours post-dose
  Area under the plasma concentration versus time curve (AUC) from Time 0 to 30 minutes post-dose (AUC0-30min), AUC from Time 0 to 12 hours post-dose (AUC0-12h), AUC from Time 0 to 24 hours post-dose (AUC0-24h), AUC from Time 0 to 96 hours post-dose (AUC0-96h), AUC from Time 0 to time of last quantifiable concentration (AUC0-t), AUC from Time 0 to infinity (AUC0-∞)
Pharmacokinetic variables in plasma in HVs only (Part I): Maximum concentration (Cmax) | Day1: from pre-dose until 96 hours post-dose
Pharmacokinetic variables in plasma in HVs only (Part I): Time to maximum concentration (tmax) | Day1: from pre-dose until 96 hours post-dose
Pharmacokinetic variables in plasma in HVs only (Part I): Terminal half-life (t½) | Day 1: from pre-dose until 96 hours post-dose
Pharmacokinetic variables in plasma in HVs only (Part I): Clearance (CL/F) | Day 1: from pre-dose until 96 hours post-dose
Pharmacokinetic variables in plasma in HVs only (Part I): Apparent volume of distribution during the terminal phase (Vz/F) | Day 1: from pre-dose until 96 hours post-dose
Pharmacokinetics variables in plasma in BE subjects (Part II); in terms of Area Under the Curve | At Day1 and 27: from pre-dose until 8 hours post-dose
  Day1: AUC0-30min, AUC0-8h, AUC0-t
  - Day27: AUC0-30min at steady state (AUC0-30min,ss), AUC0-8h at steady state (AUC0-8h,ss), AUC0-t at steady state (AUC0-t,ss)
Pharmacokinetics variables in plasma in BE subjects (Part II): Cmax | At Day1 and 27: from pre-dose until 8 hours post-dose
  Day1: Cmax
  - Day27: Cmax at steady state (Cmax,ss)
Pharmacokinetics variables in plasma in BE subjects (Part II): tmax | At Day 1 and 27: from pre-dose until 8 hours post-dose
  Day 1: tmax
  - Day27: tmax at steady state (tmax,ss)
Pharmacokinetics variables in plasma in BE subjects (Part II): Ratio of accumulation (Rac) for Cmax and AUC parameters | At Day 1 and 27: from pre-dose until 8 hours post-dose
CHF6333 plasma concentrations (Part II) | At Day 27 and 28: 3 hours post-dose
  CHF6333 plasma concentrations on Day27 and 28 will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: James D. Chalmers, Principal Investigator — School of Medicine, University of Dundee, UK
Locations (9):
- United Kingdom (9):
  - Royal Papworth Hospital NHS Foundation Trust, Cambridge Centre for Lung Infection, Cambridge
  - Tayside Medical Science Centre, Ninewells Hospital & Medical School, Dundee
  - NHS Lothian, Edinburgh
  - Glasgow Royal Infirmary, Glasgow
  - The Leeds Teaching Hospitals NHS Trust, Saint James's University Hospital, Leeds
  - Royal Bromptom Hospital (NHS Guy's and Thomas'), London
  - Manchester University NHS Foundation Trust, Manchester
  - Medicines Evaluation Unit (MEU), Manchester
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No